CLINICAL TRIAL: NCT05578222
Title: Efficacy and Safety of Pembrolizumab as First-line Treatment for Advanced Non-small Cell Lung Cancer Complicated With Chronic Obstructive Pulmonary Disease: a Prospective, Single-arm, Single-center Phase II Trial
Brief Title: Pembrolizumab as First-line Treatment for Advanced NSCLC Complicated With COPD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Chest Hospital (Other)
Responsible Party: Principal Investigator, Jianwen Qin, chief physicians, Tianjin Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSCLC+COPD-Pembrolizumab-001
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: NSCLC With COPD
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): All patients who met the inclusion criteria and did not meet the exclusion criteria were enrolled in the treatment group
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab, 200mg i.v. gtt,D1,Q3W,
  Other Names: Keytruda,NSCLC,COPD

SUMMARY:
This clinical trial aims to evaluate the efficacy and safety of pembrolizumab in the first-line treatment of advanced NSCLC complicated with COPD and its influence on the course of COPD, so as to provide prospective clinical evidence for immunotherapy of NSCLC complicated with COPD in China and to guide clinical application.

DETAILED DESCRIPTION:
This clinical study mainly includes 3 stages of screening, treatment and follow-up.

Pabolivizumab at a fixed dose of 200 mg intravenous infusion on day 1 for Q3W, continued to maintain administration for no more than 35 cycles, or until the imaging proves the early termination of PD or other protocols. Imaging evaluation is performed every 6 weeks within 6 months from the first dose of pabolizumab and approximately every 12 weeks thereafter until disease progression or early withdrawal. Conduct regular safety assessments, document changes in COPD condition, track adverse events until remission or stabilization, or restore baseline levels, or receive other anti-tumor therapy; Record the combined medications.

Main research objectives:Evaluation of PFS in patients with advanced NSCLC and COPD treatment of pabolivizumab.

Secondary research objectives:To assess the ORR and acute exacerbation rate (times/person/year) and adverse reactions of PABLIZUMAB in patients with advanced NSCLC with COPD.

Purpose of exploratory research:The expression levels of PD-L1, CD4+ and CD8+ T lymphocytes in tumor tissues of patients with NSCLC and COPD before treatment were laboratory tested, and the correlation between different COPD grades and immune cell infiltration and efficacy was explored. This study was designed as a single-armed, single-center, prospective, phase II clinical study with 30 clinical, radiographic, pulmonary function and pathologically confirmed advanced (stage IV) NSCLC combined with COPD primary treatment subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent before enrollment;
2. Men and women aged 18-75;
3. The patient must be able to provide fresh or archived tumor tissue and its pathology report;
4. No previous antitumor therapy, life expectancy is not less than 12 weeks;
5. Newly diagnosed NSCLC subjects confirmed by pathology and imaging; Stage: cT1-4N1-3M1 (stage Ⅳ), AJCC eighth edition clinical staging of lung cancer;
6. Asymptomatic patients with NSCLC brain metastases
7. PD-L1 tumor fraction (TPS) ≥1%;
8. Epidermal growth factor receptor (EGFR) gene mutation negative and anaplastic lymphoma kinase (ALK) negative;
9. Measurable lesions that meet RECIST v1.1 criteria;
10. Patients with COPD who met the relevant diagnostic criteria for COPD in the Guidelines for the Diagnosis and Treatment of Chronic Obstructive Pulmonary Disease (Revised 2021) formulated by Chinese Society of Respiratory Medicine, and whose condition was stable for ≥2 weeks;
11. ECOG PS: 0 ~ 2;
12. The functions of vital organs meet the following requirements (excluding the use of any blood components and cell growth factors within 14 days) :

    Normal bone marrow reserve, neutrophil (ANC) ≥1,500/mm³, platelet count (PLT) ≥100,000/mm³, hemoglobin (Hb) ≥5.6 mmol/L (9g/dL);Creatinine (Cr) ≤1.5 mg/d and/or Clearance of creatinine (CCr) ≥60 ml/min;Normal liver function or Total Bilirubin (TBIL) ≤1.5 ULN,Aspartate Transaminase (AST) and Alanine Transaminase (ALT) ≤1.5 ULN;
13. Non-surgical sterilization or use of a medically approved contraceptive method (e.g. intrauterine device, birth control pill, or condom) during the study treatment period and for 3 months after the end of the study treatment period;Patients with non-surgical sterilization or women of childbearing age had to have a negative serum or urine HCG test within 7 days before study enrollment; must be non-lactation period;Male patients who are not surgically sterilized or of childbearing age are required to consent to use a medically approved contraceptive method with their spouse during the study treatment period and for 3 months after the study treatment period;
14. Subjects volunteered to join this study, with good compliance, safety and survival follow-up.

Exclusion Criteria:

1. Previous radiotherapy, chemotherapy, long-term or high-dose hormone therapy, surgery, or molecular targeted therapy;
2. The subject has previous or concurrent other malignant tumors;
3. History of asthma or other respiratory diseases (bronchiectasis, tuberculosis, interstitial pneumonia, occupational lung disease, sarcoidosis, etc.);Patients with objective evidence of radiation pneumonitis, drug-associated pneumonitis, or severe impairment of pulmonary function;
4. History of lobectomy;
5. A history of clinically significant circulatory failure;
6. Significant contraindications for spirometry (history of myocardial infarction, cerebral artery or aortic aneurysm, history of eye surgery, hemoptysis);
7. Patients with rheumatic diseases;Patients with heart, cerebrovascular, liver, kidney, hematopoietic system and other serious primary diseases.
8. Patients with a history of acute gastrointestinal bleeding within 3 months;
9. Previous immune checkpoint inhibitor therapy;The subject is known to have a previous allergy to macromolecular protein preparations, or to any PD-1 mab component;
10. The subject has any active autoimmune disease or a history of autoimmune disease (e.g., but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism;Subjects with vitiligo or complete remission of asthma in childhood without any intervention as adults were included;Subjects with asthma requiring medical intervention with bronchodilators were excluded);
11. The subject has active infection or unexplained fever >38.5 ℃ during the screening period or before the first administration;
12. Subjects with innate or acquired immune deficiency, such as HIV infection, or active hepatitis (transaminases did not meet the inclusion criteria, hepatitis B reference: HBV DNA≥10⁴/ml;HCV RNA≥10³/ml);Chronic hepatitis B virus carriers, HBV DNA≥2000 IU/ml (≥10⁴ copies/ml), must receive antiviral therapy during the trial to be enrolled;
13. The subject is participating in another clinical study or it has been less than one month since the end of the previous clinical study;Subjects may receive other systemic antitumor therapy during the study;
14. Receive live vaccine less than 4 weeks before or possibly during the study period;
15. The subject cannot or does not agree to pay for the examination and treatment expenses at his own expense;
16. Pregnant or lactating women;
17. Other conditions that should be excluded from the study in the opinion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-10 (Estimated); Primary Completion 2023-12-12 (Estimated); Study Completion 2024-12-12 (Estimated)

PRIMARY OUTCOMES:
PFS | 30 months
  The time from the beginning of randomization to the progression of tumor development or death for any reason.

SECONDARY OUTCOMES:
ORR | 12 months
  The proportion of patients whose tumor volume has decreased to a prespecified value and can maintain a minimum time limit.ORR=PR+CR
Rate of acute exacerbations of COPD (times/year) | 30 months
  Acute exacerbations of COPD are coughs, sputum production, worsening of dyspnea, or increased amount of sputum, or yellow phlegm, requiring a change in medication regimen.Acute exacerbations of COPD are classified as Grades I.-III according to clinical signs.
adverse events | 30 months
  Harmful reactions that are not related to the purpose of medication under normal dosage of qualified drugs. Refer to CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: JianWen Qin, Study Director — No. 261, Taierzhuang South Road, Jinnan District, Tianjin, Tianjin Chest Hospital.
Locations (1):
- Tianjin Chest Hospital, Tianjin, China

REFERENCES:
- [Derived] Dong W, Yin Y, Liu B, Jiang Y, Wang L, Shi D, Qin J. Efficacy and safety of pembrolizumab as first-line treatment for advanced non-small cell lung cancer complicated with chronic obstructive pulmonary disease: protocol for a prospective, single-arm, single-center, phase II clinical trial. Front Oncol. 2024 Mar 7;14:1179232. doi: 10.3389/fonc.2024.1179232. eCollection 2024. PMID 38515570